CLINICAL TRIAL: NCT02959684
Title: Strategic Screening for Infectious Diseases (Tuberculosis, HIV, HBV, HCV) Amongst Migrants in France
Acronym: STRADA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Paris 7 - Denis Diderot (Other)
Responsible Party: Principal Investigator, Dr Martin Duracinsky, Dr, University Paris 7 - Denis Diderot
Other Study IDs: PROunit-STRADA2016
Record Dates: First submitted 2016-10-26; First posted 2016-11-09 (Estimated); Last update posted 2018-05-03 (Actual); Status verified 2018-05

CONDITIONS: HIV; Hepatitis C; Hepatitis B; Tuberculosis
MeSH Terms: conditions — Hepatitis C; Hepatitis B; Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To evaluate the efficacy of a new screening for infectious diseases: tuberculosis, HIV, HBV and HCV, based on risk factors questionnaires (TB screen for tuberculosis and TROD screen for HIV and hepatitis) amongst a population of legal migrants during their mandatory medical check-up. This study aims for a global improvement of screening and care for migrants.

DETAILED DESCRIPTION:
In France, the prevalence of infectious diseases such as tuberculosis, HIV/HBV/HCV is high amongst migrants originating from certain countries, hence the official guidelines recommending targeted testing. The rapid testing devices (TROD) give immediate results and reduce missed opportunities. However their use is not yet widespread and migrant populations remain insufficiently tested. Regarding the UNAIDS 90-90-90 goal, France is failing the screening part of the treatment cascade, while 90% of patients are treated and have undetectable viral load. Risk scores based on the best known risk factors for these infections (HIV/HBV/HCV) have previously been developed. They have helped build a pilot of a new unique questionnaire: TROD screen. An electronic survey, called TB screen, was designed to screen for tuberculosis amongst asylum seekers in Switzerland and validated. This survey enables to detect signs of active tuberculosis and may replace the use of pulmonary radiography, thus reducing exposure to X-rays.

It is a prospective multi-centric observational study validating screening tests for HIV/HBV/HCV in two phases:

* Phase 1: a risk score will be validated, including a qualitative study analyzing its acceptability
* Phase 2: its performance will be compared with that of a screening targeted based on the country of origin The phase 1 and phase 2 will include respectively 10.000 and 5000 participants.

For tuberculosis, the efficacy of the improved version of TB screen will be compared with a systematic radiography.

Participation to this study will be voluntary and independent from the delivery of a residence permit. Participants will be informed of it and will systematically receive information about prevention of those infectious diseases.

ELIGIBILITY:
Inclusion Criteria:

* Migrants undergoing the routine medical visit
* Giving informed consent (oral consent)

Exclusion Criteria:

* Asylum seekers
* Persons not understanding the questionnaire
* Persons aware of their HIV, HBV or HCV positive status

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Migrants undergoing the routine immigration medical visit
Sampling Method: Non-Probability Sample
Enrollment: 70000 (Estimated)
Dates: Start 2017-04-14 (Actual); Primary Completion 2018-07 (Estimated); Study Completion 2019-07 (Estimated)

PRIMARY OUTCOMES:
Comparison of the number of HIV, HBV or HCV positive patients identified in both arms of the screening strategy. | 2 years
Number of tuberculosis patients identified through the modified TB screen questionnaire | 2 years

SECONDARY OUTCOMES:
Number of HIV/HBV/HCV patients linked to care after being identified through TROD screen. | 2 years
Predictive value of the questionnaire TROD screen. | 2 years
Predictive value of the questionnaire TB screen. | 2 years
Cost-effectiveness of the TROD screen questionnaire compared with a non-targeted screening, calculated in terms of cost per QALY (quality-adjusted life years) gained through this program | 2 years

CONTACTS AND LOCATIONS:
Locations (18):
- France (18):
  - OFII Bordeaux, Bordeaux
  - OFII Cergy, Cergy
  - OFII Clermont-Ferrand, Clermont-Ferrand
  - OFII Grenoble, Grenoble
  - OFII Lille, Lille
  - OFII Lyon, Lyon
  - OFII Marseille, Marseille
  - OFII Melun, Melun
  - OFII Metz, Metz
  - OFII Montpellier, Montpellier
  - OFII Montrouge, Montrouge
  - OFII Nantes, Nantes
  - OFII Nice, Nice
  - OFII Orléans, Orléans
  - OFII Reims, Reims
  - OFII Rennes, Rennes
  - OFII Rouen, Rouen
  - OFII Toulouse, Toulouse

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Meffre C, Le Strat Y, Delarocque-Astagneau E, Dubois F, Antona D, Lemasson JM, Warszawski J, Steinmetz J, Coste D, Meyer JF, Leiser S, Giordanella JP, Gueguen R, Desenclos JC. Prevalence of hepatitis B and hepatitis C virus infections in France in 2004: social factors are important predictors after adjusting for known risk factors. J Med Virol. 2010 Apr;82(4):546-55. doi: 10.1002/jmv.21734. PMID 20166185
- [Background] Schneeberger Geisler S, Helbling P, Zellweger JP, Altpeter ES. Screening for tuberculosis in asylum seekers: comparison of chest radiography with an interview-based system. Int J Tuberc Lung Dis. 2010 Nov;14(11):1388-94. PMID 20937177
- [Background] d'Almeida KW, Kierzek G, de Truchis P, Le Vu S, Pateron D, Renaud B, Semaille C, Bousquet V, Simon F, Guillemot D, Lert F, Cremieux AC; Emergency Department HIV-Screening Group. Modest public health impact of nontargeted human immunodeficiency virus screening in 29 emergency departments. Arch Intern Med. 2012 Jan 9;172(1):12-20. doi: 10.1001/archinternmed.2011.535. Epub 2011 Oct 24. PMID 22025095
- [Background] d'Almeida KW, Pateron D, Kierzek G, Renaud B, Semaille C, de Truchis P, Simon F, Leblanc J, Lert F, Le Vu S, Cremieux AC. Understanding providers' offering and patients' acceptance of HIV screening in emergency departments: a multilevel analysis. ANRS 95008, Paris, France. PLoS One. 2013 Apr 29;8(4):e62686. doi: 10.1371/journal.pone.0062686. Print 2013. PMID 23638133
- [Background] Bottero J, Boyd A, Gozlan J, Carrat F, Nau J, Pauti MD, Rougier H, Girard PM, Lacombe K. Simultaneous Human Immunodeficiency Virus-Hepatitis B-Hepatitis C Point-of-Care Tests Improve Outcomes in Linkage-to-Care: Results of a Randomized Control Trial in Persons Without Healthcare Coverage. Open Forum Infect Dis. 2015 Oct 26;2(4):ofv162. doi: 10.1093/ofid/ofv162. eCollection 2015 Dec. PMID 26668814
- [Background] Haukoos JS, Lyons MS, Lindsell CJ, Hopkins E, Bender B, Rothman RE, Hsieh YH, Maclaren LA, Thrun MW, Sasson C, Byyny RL. Derivation and validation of the Denver Human Immunodeficiency Virus (HIV) risk score for targeted HIV screening. Am J Epidemiol. 2012 Apr 15;175(8):838-46. doi: 10.1093/aje/kwr389. Epub 2012 Mar 19. PMID 22431561
- [Derived] Duracinsky M, Yaya I, Yombo-Kokule L, Bessonneau P, Thonon F, Rousset-Torrente O, Roudot-Thoraval F, Lert F, Zucman D, Chassany O. Development of a risk prediction score for screening for HBV, HCV and HIV among migrants in France: results from a multicentre observational study (STRADA study). BMJ Open. 2024 Jun 5;14(6):e075315. doi: 10.1136/bmjopen-2023-075315. PMID 38839381